CLINICAL TRIAL: NCT01443754
Title: Hybrid Revascularisation by Combined CABG and PCI in Multivessel Coronary Disease. An Observational Study.
Brief Title: Hybrid Revascularisation by Combined Coronary Artery Bypass Graft (CABG) and PCI in Multivessel Coronary Disease
Acronym: HYBRID
Status: Terminated | Type: Observational
Why Stopped: Lack of recruitment
Sponsor: Ettore Sansavini Health Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ESREFO04
Record Dates: First submitted 2011-09-20; First posted 2011-09-30 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2015-02

CONDITIONS: Coronary Artery Disease (CAD)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hybrid group: Patients with multi-vessel coronary artery disease (CAD) amenable to hybrid revascularization (LIMA-LAD surgical revascularization followed by PCI)
  Interventions: Procedure: LIMA-LAD surgical revascularization; Procedure: PCI

INTERVENTIONS:
Procedure: LIMA-LAD surgical revascularization — Off-pump coronary artery bypass (OPCAB) in which coronary revascularization is performed on the beating heart will be followed, the choice of the technical solutions being left at the discretion of the cardiac surgeon:
  * use of a left anterior small thoracotomy (LAST), LIMA harvesting using thoracoscopic methods and manual anastomosis of the LIMA-LAD using a stabilization device;
  * minimally invasive direct coronary bypass surgery (MIDCAB). The procedures can be performed alone or in combination with one another.
Procedure: PCI — State of the art drug eluting stent (DES)-based percutaneous coronary intervention will be used by each participating site, according to current international guidelines.
  Zotarolimus, everolimus or sirolimus drug-eluting stents will be used in all sites.

SUMMARY:
The present study is designed as a prospective, single centre, open label, observational trial.

The study will collect information about the medical care patients receive during their planned procedure(s). No new testing or procedures will be done.

Patients elected for hybrid revascularization will be asked their written consent to the use of their personal data.

Left internal mammary artery to the Left Anterior Descending Coronary Artery (LIMA-LAD)surgical revascularization will be performed first, followed by percutaneous revascularization of the other vessels in the frame of the same hospitalization.

After discharge patients will attend clinic visits at 30 days and 12 months, as per usual clinical practice, and will be contacted by phone at 6 months after procedure. Angiographic follow-up will be performed in symptomatic patients, as clinically indicated.

DETAILED DESCRIPTION:
Hybrid coronary revascularization integrates the positive features of both Percutaneous Coronary Intervention (PCI) and Coronary Artery Bypass Graft (CABG), combining the durability of Left Anterior Descending Coronary Artery (LIMA) coronary bypass with the minimal invasiveness and lower risk of percutaneous intervention. Thereby it might represent a better option in a sizeable proportion of patients.

Candidate patients in whom hybrid revascularization would be advantageous are several subgroups of Coronary Artery Disease (CAD) patients that are increasing in numbers: the elderly patients with a high risk of mortality and/or morbidity for CABG, patients with significant disabilities and patients in whom treatment durability is important but a significantly invasive approach is not an option.

There are several potential advantages of the hybrid procedure over conventional CABG in selected patients. These advantages include the avoidance of cardiopulmonary bypass-related morbidity, no aortic manipulation with the LIMA-LAD with the beating heart procedure, less blood loss and decreased transfusions, a shorter recovery time than after conventional CABG and patient's preference for "minimally invasive" surgery.

The investigators hypothesize that in selected patients with diffuse coronary disease, a "hybrid" approach employing a staged revascularisation procedure may allow to lower the surgical risk, increase the completeness and effectiveness of revascularisation and, hopefully, to improve immediate and long term outcome.

To test this hypothesis, a well designed, properly sized, prospective, randomized study is needed. Available data, however, do not provide sufficient information to speculate on a clinically meaningful, yet achievable, effectiveness.

Aim of this observational study is therefore to collect more information on the target population, the clinical outcomes and optimal management in order to inform the design of a comparative effectiveness trial.

ELIGIBILITY:
Inclusion Criteria:

Patients with multi-vessel coronary artery disease (CAD) amenable to hybrid revascularization and fulfilling the following criteria:

1. ≥70% left-anterior descendent (LAD) obstruction suitable for surgical revascularization using the left internal mammary artery (LIMA);
2. patients amenable to a off-pump beating heart revascularization procedure;
3. non-LAD coronary lesions suitable for percutaneous coronary artery intervention (PCI), as adjudicated by one interventional cardiologist and one cardiac surgeon;
4. ≥ 70 years of age
5. Written informed consent for the use of personal data

Exclusion Criteria:

1. patients hemodynamically unstable;
2. acute or recent (< 1 month) myocardial infarction;
3. severe heart failure (NYHA Class IV);
4. creatinine > 2.2 mg/dl;
5. allergy to radiographic contrast;
6. contraindication to double antiaggregation therapy (DAT) for at least 12 months;
7. previous cardiac surgery of any type;
8. previous thoracic surgery involving left pleural space;
9. previous coronary stenting: within one month for BMS, within 6 months for DES;
10. disabling stroke within previous 6 months;
11. need for concomitant cardiac surgery during index hospitalization;

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients referred to participating sites with clinical indication to revascularization and with clinical characteristics and multi-vessel disease amenable to hybrid revascularization
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
composite of major cardiac and cerebrovascular events (MACCE) | From date of inclusion until the date of first documented MACCE, assessed up to 12 months
  composite of major cardiac and cerebrovascular events, i.e. the first occurrence of any of the following events:
  * Death from any cause
    * From cardiovascular causes
    * From noncardiovascular causes
  * Stroke
  * MI
  * hospitalization for repeat revascularization procedure

SECONDARY OUTCOMES:
• Procedural success | during index hospitalization up to discharge from the hospital ( expected average of hospital stay: 2 weeks)
  successful treatment will be declared when a complete hybrid revascularisation in the absence of complications during the index hospitalization has been achieved.
• Procedural and post-procedural blood loss and number of transfusions | during index hospitalization up to discharge from the hospital ( expected average of hospital stay: 2 weeks)
• Recovery time | from end of intervention up to discharge from the hospital (expected average of hospital stay: 2 weeks)
  time to extubation; number of days in ICU; total duration of hospital admission
• New York Heart Association (NYHA) class modification with respect to baseline | at 12 months post-procedure
Quality of life (SF-12 questionnaire) | at 12 months post-procedure
Length of time to return to work or normal activities | from hospital discharge (index hospitalization) up to date of return to work or normal activities assessed up to 12 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Del Giglio, MD, Principal Investigator — GVM Care & Research
Locations (1):
- Maria Cecilia Hospital, Cotignola, Ravenna, Italy

IPD SHARING:
Plan to Share IPD: No